CLINICAL TRIAL: NCT02300818
Title: Magneto Therapy in the Therapy of Glaucoma
Brief Title: Effects of Magnetic Therapy and Seawater Combined in Decreasing Intraocular Presion.
Acronym: GME
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American Society Of Thermalism And Climatology Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20141110
Record Dates: First submitted 2014-11-14; First posted 2014-11-25 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Primary Open Angle Glaucoma; Hypertension Ocular
Keywords: Hipertension ocular, Glaucoma, Magnetotherapy, seawater
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulsed Electromagnetic Field Therapy (Active Comparator): Pulsed Electromagnetic Field Therapy widely termed as (PEMF) is a reparative technique used for treatment of eye therapy has proved to be a beneficial treatment for those suffering from glaucoma. This therapy helps in increased blood flow and show positive results on latent, initial and advanced glaucoma with ten sessions of seven minutes' each.
  PEMF has also proved to be beneficial in vision acuity of patients with low vision. In 50 per cent of the cases, values improved. Patients with vision acuity of 0.2 diopters showed improvement from 46 before treatment to 75 after treatment.
  Different studies on varied diseases have proved that Pulsed Electromagnetic Field Therapy (PEMF) treatment is a safe, non-invasive and effective option for curing ocular conditions.
  Interventions: Device: Pulsed Electromagnetic Field Therapy
- Seawater eyedrops (Active Comparator): instantly soothes and clears the eye irritation caused by pollution, pollen, smoke, etc. It is a very practical system for eye daily hygiene · enables efficient therapeutic help in basic eye conditions such as: · · internal and external stye blepharitis and keratoconjunctivitis · · Conjuntiviti Episcleritis and scleritis
  Interventions: Drug: Seawater eyedrops

INTERVENTIONS:
Device: Pulsed Electromagnetic Field Therapy — Pulsed Electromagnetic Field Therapy widely termed as (PEMF) is a reparative technique used for treatment of eye therapy has proved to be a beneficial treatment for those suffering from glaucoma. This therapy helps in increased blood flow and show positive results on latent, initial and advanced glaucoma with ten sessions of seven minutes' each.
  Other Names: Field magnetic in Glaucoma
  Arms: Pulsed Electromagnetic Field Therapy
Drug: Seawater eyedrops — Eye-drops daily 1 time a day for 12 weeks
  Other Names: thalassotherapy ocular
  Arms: Seawater eyedrops

SUMMARY:
Glaucoma is among the leading causes for blindness in the western world. Elevated intraocular pressure (IOP) has been identified as the most important risk factor. However, some patients progress despite adequate IOP lowering while some subjects with elevated IOP never develop glaucoma. Other patients develop glaucoma although IOP measurements were always in the normal range. Therefore, other factors must be involved. In the last years, studies using MRI have been performed and evidence has accumulated that also changes in retrobulbar structures are present, in particular in the lateral geniculate nucleus and the visual cortex. However, these studies were limited by the low spatial resolution of the MRI instruments used.

DETAILED DESCRIPTION:
The two principal pathophysiological mechanisms of glaucomatous process (hydromechanical and metabolic) determine the development of two trends in the treatment of glaucoma. One treatment modality is aimed at reduction of intraocular pressure, the other at therapy of hemodynamic and metabolic disorders. General and local drug therapy and physiotherapy, including electro- and laser stimulation of the retina and optic nerve and magneto-therapy, are used to correct these disorders. Modern ocular hypotensive agents are myotics and beta-adrenoblockers, adrenergic drugs, alpha 2-agonists, carboanhydrase inhibitors, some prostaglandins, osmotic agents. The progress attained in conservative therapy of glaucoma should by no means be overstated. In many cases only a combination of conservative and surgical methods of treatment helps preserve vision in a glaucoma patient.

During the following investigation we will demonstrate that the use of Magneto therapy Ocular (MTO) reverses the symptomatology in Glaucoma patients. The use of Eyeglass magnetic prevents the development of Glaucoma disease.During the following investigation we will demonstrate that the use of MTO reverses the symptomatology of Glaucoma patients; the use of seawater as drops prevents the development of Glaucoma disease and the combined use of MTO and seawater is an effective therapy against Glaucoma disease that will cure a grand percentage of the patients.

We will randomized 100 glaucoma patients and will treat them with MTO (group 1) and seawater drop (group 2) and combined group 3 and will compare results

ELIGIBILITY:
Inclusion Criteria:

Patient is aged 18 years or older, with glaucoma include poorly controlled open angle glaucoma (Pigmentary & Exfoliative Glaucoma) Patient is willing to participate in the 3-month study and to adhere to the follow-up schedule.

Patient is willing to review and sign a consent form.

Exclusion Criteria:

Prior glaucoma surgery other than laser trabeculoplasty or peripheral iridotomy.

Patient has mental impairment such that he/she could not understand the protocol or is not in a position to provide written informed consent.

Patient is pregnant. Patient might require other ocular surgery within the 6-month follow-up period. Having concurrent treatment with systemic steroids. Patient is under 18 years old -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Intro-ocular pression after magnetic field exposition | 12 weeks
  Pulsed Electromagnetic Field Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Garis Silega, Principal Investigator — America Society of thermalism
Locations (1):
- Gaviota Clinic, Newark, New Jersey, United States